CLINICAL TRIAL: NCT07358104
Title: Investigating the Efficacy of Camel Whey Protein and Camel Whey Protein Nanoparticles for Treating Intra-bony Periodontal Defects: Randomized Clinical Trial
Brief Title: Efficacy of Camel Whey Protein and Camel Whey Protein Nanoparticles for Treating Intra-bony Periodontal Defects
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Walid Elamrousy, Professor and postgrad course director of Periodontology Department Faculty of Oral and Dental Medicine,Kafrelsheikh University, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KFSIRB200-317
Record Dates: First submitted 2026-01-02; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Periodontal Diseases; Periodontal Attachment Loss
MeSH Terms: conditions — Periodontal Diseases; Periodontal Attachment Loss

STUDY DESIGN:
Intervention Model Description: healthy patients with Stage III or IV periodontitis will be selected from the outpatient clinic of the Department of Periodontology, sulcular incisions will be performed followed by elevation of mucoperiosteal flaps and granulation tissue curettage then various interventions will be applied to each group
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: participant , investigator and outcome assessors are masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Open currettage (Experimental): open flap debridement
  Interventions: Drug: only open flap debridement
- Open curettage with scaffold material (Placebo Comparator): scaffold material
  Interventions: Drug: scaffold material
- Open curettage with Camel whey protein (Active Comparator): CWP
  Interventions: Drug: CWP
- Open curettage with Camel whey protein nanoparticle (Active Comparator): CWP NPs
  Interventions: Drug: CWP NPs

INTERVENTIONS:
Drug: only open flap debridement — only open flap granulation tissue debridement
  Arms: Open currettage
Drug: scaffold material — open flap debridement with defect filling with scaffold material
  Arms: Open curettage with scaffold material
Drug: CWP — open flap debridement with defect filling with CWP
  Arms: Open curettage with Camel whey protein
Drug: CWP NPs — open flap debridement with defect filling with CWP NPs
  Arms: Open curettage with Camel whey protein nanoparticle

SUMMARY:
Intraosseous bone defects (IOBDs) are a significant challenge in the treatment of periodontal disease. Several bone graft materials can be used for bone defect regeneration.

Camel whey protein (CWP) has emerged as a promising alternative due to its unique properties, including: High biological value containing essential amino acids, anti-inflammatory, antioxidant and immunomodulatory effects.

However, the therapeutic application of CWP for bone regeneration can be limited by its solubility and bioavailability . Nanoparticles offer a novel approach to enhance drug delivery and improve therapeutic efficacy. Introduction of bone grafts in the form of nanoparticles was found to improve the bioactivity and biocompatibility of artificial bone graft.

Nanoparticles (NPs) can efficiently enter biological organisms due to their very tiny size. The ability of NPs to easily pass through even the smallest blood capillaries and escape being phagocytized due to their small size (1-100 nm) extends their plasma half-life and permits a more progressive release of the medication. Nanoparticles have quicker absorption and a relatively greater drug loading arise from interactions at the surface. NPs increased antibacterial action may be attributed to their huge surface area and high charge density, which allows them to interact with the negatively charged surface of bacterial cells

DETAILED DESCRIPTION:
Periodontitis is clinically characterized by loss of gingival tissue attachment to the tooth, deepening of periodontal pocket, degradation of the periodontal ligament, and loss of alveolar bone. This destructive process is associated with the presence of subgingival microbial communities and dense immuno-inflammatory infiltrate in the periodontium that may lead to tooth loss if not appropriately treated.

Periodontitis is associated with a dysbiotic polymicrobial community, in which different members have distinct and synergistic roles that promote destructive inflammation. Inflammation, in turn, can exacerbate dysbiosis through provision of nutrients for the bacteria (derived from tissue breakdown products; eg, collagen peptides and hemecontaining compounds). Therefore, inflammation and dysbiosis are reciprocally reinforced and generate a positive-feedback loop. This self-sustaining loop may underlie the chronicity of periodontitis, the development of which requires a susceptible host.

Risk factors include the presence of bacteria that subvert the host response, systemic disease, smoking, aging and immune deficiencies. These factors could promote dysbiosis by acting individually or, more effectively, in combination.

Periodontal defects have been differentiated based on bone resorption patterns into "supraosseous" ("suprabony") and "infraosseous" ("infrabony") "). Infrabony defects are classified according to the location and number of osseous walls remaining around the pocket. According to the classification by Goldman & Cohen , inrtabony defects are categorized as follows: (i) one-wall intrabony defects: defects bounded by one osseous wall and the tooth surface; (ii) two-wall intrabony defects: defects bounded by two osseous walls and the tooth surface; (iii) three-wall intrabony defects: defects bounded by three osseous walls and the tooth surface.

It has been suggested that the term "intrabony" means "within or inside the bone", while "infrabony" means "below the crest of bone". The authors suggested that only 3-wall angular defects should be termed "intrabony", while all other vertical bony defects should be referred to as "infrabony".

Intraosseous bone defects (IOBDs) are a significant challenge in the treatment of periodontal disease. Several bone graft materials can be used for bone defect regeneration.

Camel whey protein (CWP) has emerged as a promising alternative due to its unique properties, including: High biological value containing essential amino acids, anti-inflammatory, antioxidant and immunomodulatory effects.

However, the therapeutic application of CWP for bone regeneration can be limited by its solubility and bioavailability . Nanoparticles offer a novel approach to enhance drug delivery and improve therapeutic efficacy. Introduction of bone grafts in the form of nanoparticles was found to improve the bioactivity and biocompatibility of artificial bone graft.

Nanoparticles (NPs) can efficiently enter biological organisms due to their very tiny size. The ability of NPs to easily pass through even the smallest blood capillaries and escape being phagocytized due to their small size (1-100 nm) extends their plasma half-life and permits a more progressive release of the medication. Nanoparticles have quicker absorption and a relatively greater drug loading arise from interactions at the surface. NPs increased antibacterial action may be attributed to their huge surface area and high charge density, which allows them to interact with the negatively charged surface of bacterial cells.

ELIGIBILITY:
Inclusion Criteria:

* The patient age range will be 18-45 years of both sexes Stage III or IV periodontitis (probing depth ≥ 6 mm in teeth and clinical attachment ≥ 5 mm).
* Clinical and radiographic confirmation of 3 wall intrabony defects.
* Absence of any complicating systemic condition that may contraindicate surgical procedures.
* Adequate oral hygiene.
* Eligible participants should present good general health and agree to random assignment to any of the parallel study groups.

Exclusion Criteria:

* Allergy
* Uncontrolled systematic disorders as, diabetes mellitus, uncontrolled periodontal disease, history of head and neck radiotherapy, smokers, pregnancy, noncompliant patients, uncooperative individuals or those unable to attend the study follow-up appointments.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-01-06 (Estimated); Primary Completion 2026-07-24 (Estimated); Study Completion 2026-08-04 (Estimated)

PRIMARY OUTCOMES:
bone fill | 6-months
  Radiographic bone fill will be assessed using CBCT by subtracting the preoperative and postoperative x-rays, followed by measuring the resultant bone volume in mm³.

SECONDARY OUTCOMES:
bone density | 6-months
  radiogeaphic bone density will be assessed using CBCT
Clinical probing pocket depths | 6-months
  Clinical probing pocket depths will be measured in mm from gingival margin to the base of the sulcus using graduated periodontal probe
clinical attachment level | 6-months
  clinical attachment level will be measured in mm from cementoenamel junction to the base of the sulcus using graduated periodontal probe

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry, kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
undecided